CLINICAL TRIAL: NCT00297323
Title: An Open Observational Safety Study During Administration of Topamac, as Monotherapy in Epileptic Patients With no Prior Treatment or Unsuccessfully Treated With Other Antiepileptic Drug
Brief Title: An Observational Study of the Safety of Topiramate in Adults and Children With Epilepsy
Status: Completed | Type: Observational
Sponsor: Janssen Cilag Pharmaceutica S.A.C.I., Greece (Industry)
Responsible Party: Medical Affairs Director, Janssen Cilag Pharmaceutica S.A.C.I., Greece
Other Study IDs: CR002119
Record Dates: First submitted 2006-02-24; First posted 2006-02-28 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Seizures, Epileptic
Keywords: Seizures; Epilepsy; Topiramate; Epilepsy in Children
MeSH Terms: conditions — Seizures; Epilepsy | interventions — Topiramate

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- 001
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Topiramate — 75 patients over the age of 2 years old with epilepsy.

SUMMARY:
The purpose of this observational study is to evaluate the safety of topiramate in adults and children with epilepsy (or seizures) who have not received or have not responded to treatment with previous antiepileptic medication.

DETAILED DESCRIPTION:
Topiramate is a medication that is approved for the treatment of seizures. In accordance with international guidelines, studies are conducted after a drug is marketed to continue to evaluate and expand the knowledge regarding its safety. This is a multi-center, open-label observational safety study to collect information regarding the dosage, tolerability and effectiveness of topiramate in adults and children with epilepsy (or seizures). Patients who have not received previous treatment for epilepsy or for whom previous treatment was ineffective or intolerable will receive 6 months of treatment with topiramate. Topiramate will be given at low doses initially and gradually increased as needed for each patient to control seizure activity. Safety evaluations (incidence of adverse events and laboratory tests) and assessment of patient health status will be performed throughout the study. Effectiveness will be evaluated by recording the frequency of seizures occurring during the study. Patient and physician satisfaction with topiramate treatment will also be recorded. At the end of the study, the treating physician may continue treatment with topiramate in responding patients as appropriate. The study hypothesis is that topiramate will be effective in achieving and maintaining control of seizure activity and is well-tolerated. Observational study - No investigational drug administered.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have not received previous treatment with antiepileptic medications or patients who did not respond to previous treatment with antiepileptic medications, defined as a lack of effectiveness of the medication(s), or the inability to take the medication(s) due to adverse effects

Exclusion Criteria:

* Patients not suffering from epilepsy, whose seizures are due to other causes including disease, exposure to harmful substances, active infection or tumor and are manageable
* Patients with a hypersensitivity to topiramate or to some of its components
* Patients who should not take Topiramate for reasons listed in its approved Summary of Product Characteristics (printed information about a medication that describes its actions, side effects and intended patients)
* Patients who are uncooperative or for whom obtaining compliance with study visit schedules and procedures and information required by the study would be difficult

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In this study a total number of 75 patients will be enrolled. Adults and children over 2 years of age who are eligible according to the approved SmPC of topiramate and their seizures are not manageable. Patients with new exposure to an AE treatment for epilepsy or lack of response to the previous treatment. Patients who will agree to sign the written informed consent for the anonymous and confidential use of their medical data with their participation in the study or a relative or a legal authorised representative.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2005-06; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome is efficacy. | Visit 1-5

SECONDARY OUTCOMES:
Tolerability | Visit: 1-5
Safety of topiramate monotherapy | Visit: 1-5

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Pharmaceutica S.A.C.I. Clinical Trial, Study Director — Janssen-Cilag Pharmaceutica S.A.C.I.